CLINICAL TRIAL: NCT07012954
Title: ctDNA-Guided Rechallenge With Cetuximab Plus Trifluridine/Tipiracil Versus Bevacizumab Plus Trifluridine/Tipiracil for RAS/BRAF Wild-Type Refractory Metastatic Colorectal Cancer: A Randomized Clinical Trial
Brief Title: ctDNA-Guided Cetuximab or Bevacizumab Plus Trifluridine/Tipiracil in RAS/BRAF Wild-Type mCRC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Deshen Wang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHALLENGE-CRC
Record Dates: First submitted 2025-05-24; First posted 2025-06-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Metastatic
Keywords: ctDNA profiling; RAS/BRAF wild-type mCRC; cetuximab plus trifluridine/tipiracil; bevacizumab plus trifluridine/tipiracil; rechallenge therapy
MeSH Terms: interventions — Cetuximab; trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, multicenter clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cetuximab plus trifluridine/tipiracil (Experimental): Trifluridine/tipiracil 35 mg/m² (orally for 5 days, followed by 9 days off) plus cetuximab 500 mg/m² intravenous drip (IVD) once every two weeks.
  Interventions: Drug: Cetuximab (Erbitux, C225); Drug: trifluridine/tipiracil
- bevacizumab plus trifluridine/tipiracil (Active Comparator): Trifluridine/tipiracil 35 mg/m² (orally for 5 days, followed by 9 days off) plus bevacizumab 5 mg/kg administered by intravenous drip (IVD), repeated every two weeks.
  Interventions: Drug: trifluridine/tipiracil; Drug: Bevacizumab ( Avastin)

INTERVENTIONS:
Drug: Cetuximab (Erbitux, C225) — cetuximab 500 mg/m² repeated every two weeks.
  Other Names: Erbitux; C225
  Arms: cetuximab plus trifluridine/tipiracil
Drug: trifluridine/tipiracil — Trifluridine/tipiracil 35 mg/m² (orally for 5 days, followed by 9 days off)
Drug: Bevacizumab ( Avastin) — bevacizumab 5 mg/kg
  Arms: bevacizumab plus trifluridine/tipiracil

SUMMARY:
The objective of this randomized controlled clinical trial is to evaluate the efficacy of ctDNA-guided rechallenge with cetuximab plus trifluridine/tipiracil compared with bevacizumab plus trifluridine/tipiracil in patients with treatment-refractory, RAS/BRAF wild-type metastatic colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) remains a major public health challenge in China, where its incidence and mortality continue to rise. Although surgical resection is the cornerstone of curative treatment, metastatic disease develops in 30-40% of patients. Anti-epidermal growth factor receptor (anti-EGFR) monoclonal antibodies such as cetuximab and panitumumab are pivotal therapeutic agents for patients with RAS wild-type metastatic colorectal cancer (mCRC), exerting antitumor effects through inhibition of the EGFR pathway and activation of antibody-dependent cell-mediated cytotoxicity.

Recent evidence from phase II trials and retrospective analyses has suggested that rechallenge with anti-EGFR monoclonal antibodies in later-line settings may confer clinical benefit in selected patients who previously responded to first-line anti-EGFR-based therapy. Studies such as CRICKET and CHRONOS have highlighted the feasibility of this approach, with emerging data supporting the utility of circulating tumor DNA (ctDNA) to guide patient selection based on RAS, BRAF, and EGFR extracellular domain mutation status. Notably, the VELO study demonstrated improved progression-free survival (PFS) with third line panitumumab plus trifluridine/tipiracil compared to trifluridine/tipiracil alone, particularly in patients with ctDNA-confirmed RAS/BRAF wild-type status. Similarly, the ongoing PARERE and recently reported CITRIC studies have further emphasized the value of molecular stratification using liquid biopsy to refine anti-EGFR rechallenge strategies and optimize treatment sequencing.

The current study builds upon these findings and aims to evaluate and compare the efficacy and safety of cetuximab plus trifluridine/tipiracil versus bevacizumab plus trifluridine/tipiracil as later-line treatments in Chinese patients with RAS/BRAF wild-type mCRC, with treatment selection informed by ctDNA profiling. By integrating real-world clinical data and contemporary molecular diagnostics, this study seeks to assess the potential benefit of cetuximab-based rechallenge therapy in a population with limited therapeutic options and to contribute further evidence supporting the implementation of personalized, biomarker-guided strategies in later-line mCRC management.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma
* Initial RAS/BRAF wild-type status
* Received first-line treatment with FOLFOX, FOLFIRI, or FOLFOXIRI combined with cetuximab, with documented clinical benefit (CR/PR/SD) and progression-free survival (PFS) ≥ 6 months
* Disease progression occurred during or within 3 months after cetuximab-based first-line therapy
* Experienced further tumor progression after receiving second-line or subsequent treatments
* At least 4 months have elapsed since the last administration of cetuximab
* At least one measurable lesion according to RECIST v1.1
* RAS/BRAF wild-type status confirmed by blood-based ctDNA testing
* Normal hematologic function (platelets > 90 × 10⁹/L; white blood cells > 3 × 10⁹/L; neutrophils > 1.5 × 10⁹/L; hemoglobin > 10.0 g/100 ml)
* Serum bilirubin ≤ 1.5 × upper limit of normal (ULN), transaminases ≤ 5 × ULN
* No ascites, normal coagulation function, serum albumin ≥ 35 g/L
* Child-Pugh class A liver function
* Serum creatinine below ULN or calculated creatinine clearance > 50 ml/min (using the Cockcroft-Gault formula)
* ECOG performance status of 0-1
* Expected survival > 3 months
* Signed written informed consent
* Willing and able to undergo follow-up until death, study completion, or study termination

Exclusion Criteria:

* Presence of RAS or BRAF gene mutations
* Severe arterial embolism or ascites
* Bleeding tendency or coagulation disorders
* Hypertensive crisis or hypertensive encephalopathy
* Severe and uncontrolled systemic complications such as infections or diabetes
* Clinically significant cardiovascular diseases, including cerebrovascular accident (within 6 months prior to enrollment), myocardial infarction (within 6 months prior to enrollment), uncontrolled hypertension despite appropriate medical therapy, unstable angina, congestive heart failure (NYHA class II-IV), or arrhythmias requiring medical treatment History of or physical examination indicating central nervous system diseases (e.g., primary brain tumor, epilepsy not controlled with standard therapy, any brain metastases, or history of stroke)
* History of other malignancies within the past 5 years (excluding adequately treated basal cell carcinoma of the skin, carcinoma in situ of the cervix, and/or thyroid cancer)
* Known allergy to any of the study drugs
* Pregnant or breastfeeding women
* Women of childbearing potential (within 2 years of last menstruation) or men with reproductive potential who are not using or refuse to use effective non-hormonal contraception (e.g., intrauterine device, barrier method with spermicidal gel, or sterilization)
* Inability or unwillingness to comply with the study protocol
* Any other disease, functional impairment caused by metastatic lesions, or suspicious findings on physical examination that may indicate contraindications to study treatment or place the patient at high risk of treatment-related complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Assessed after every 4 cycles (each cycle is 14 days) from treatment initiation until radiographic disease progression, treatment discontinuation, or completion of the 5-year follow-up, whichever occurs first
  The percentage of patients in a study group who have a partial or complete response to treatment according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
Progression Free Survival | Assessed throughout the study duration (5 years)
  The proportion of patients who remain alive and whose disease does not progress after starting treatment
Overall survival | Assessed throughout the study duration (5 years)
  Time from treatment initiation to death from any cause or censored due to loss to follow up
Adverse events | Assessed throughout the study duration (5 years)
  Assessment of adverse events and their severity according to NCI CTCAE version 5.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Data and materials used in this study can be made available following study completion upon reasonable request to the corresponding author, subject to ethical and legal considerations and applicable data-sharing agreements.